CLINICAL TRIAL: NCT00814190
Title: Effect of Internet Therapeutic Intervention on A1C Levels in Type 2 Diabetes Mellitus
Brief Title: Effect of Internet Therapeutic Intervention on A1C Levels in Type 2 Diabetes Mellitus (DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrine Research Society (Other)
Responsible Party: Dr. Hugh Tildesley, Providence Health Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Internet Intervention in T2D
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Internet Therapeutic Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Intervention (Experimental): The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Interventions: Other: Internet Intervention
- Standard Care (No Intervention): This arm will receive standard care which includes self-blood glucose monitoring at least 3 times daily and visit to the endocrinologist at least once every 3 months.

INTERVENTIONS:
Other: Internet Intervention — The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Other Names: Remote Glucose Monitoring System
  Arms: Internet Intervention

SUMMARY:
Management of diabetes is an evolving challenge to health care professionals. The fluctuations of glucose levels over the lifetime of patients with diabetes can lead to complications such as nephropathy, neuropathy, retinopathy and cardiovascular diseases. Although diabetes is a chronic disease, it can be controlled with use of medications (pills or insulin), and/or changes in life-style and diet. These interventions are aimed at keeping the blood glucose levels normal or in the range of acceptable levels.

An important aspect of diabetes care is the monitoring of blood glucose levels in order to assess the effectiveness of treatment and to modify the treatment to achieve the desirable glucose levels. Patients with type 2 DM treated with insulin are recommended to perform testing for their blood glucose levels; however, it often requires intervention by health professionals in order to prevent the immediate and serious complications of hyper or hypoglycemia. The frequent self-monitoring of blood glucose and effective interventions by the health professionals may eventually allow tighter control of blood glucose levels and delay or prevent the complications associated with diabetes.

In this study, the investigators wish to evaluate the effect of an Internet based remote monitoring system that allows for patients to upload their blood glucose readings online and for the health care professional to view and provide feedback or therapeutic intervention. The Internet based system has the features of presenting the blood glucose readings according to the time of day and automatically calculates the daily average plus the standard deviation. A visual graph of the glucose readings over a 24-hour period is also generated for view. In addition, the doctor can give feedback by sending messages through the system. The patient's personal information is kept secure as outlined by the privacy policy of the Internet based system and only the doctor and the patient can view the uploaded glucose readings.

The investigators propose that the standardized encounters using the Internet will improve the outcome of treatment for patients with type 2 DM.

DETAILED DESCRIPTION:
Purpose: To determine whether use of an Internet-based glucose monitoring system improves A1C levels in patients with type 2 diabetes mellitus.

Hypothesis:We propose that the standardized encounters between the patient and the health care profession using the Internet will improve the outcome of treatment for patients with type 2 DM.

Justification:The standard treatment will involve glucose monitoring by testing blood glucose 3 times daily, performing a laboratory test of blood hemoglobin every three months, and visiting the doctor every three months for standard care. All of the subjects will be under standard care; however, half will also use the Internet system to report glucose readings which will allow the health care professional to view the results and to provide feedback.

Research Method: Type 2 diabetes patients who satisfy the inclusion criteria will be recruited from St. Paul's Diabetes Teaching and Training Centre. They will be randomized into 2 groups (Intervention and Control). There is an equal chance, a 50/50 chance, of being placed in either group. The control subject group will receive standard care and will be asked to perform self-blood glucose monitoring 3 times daily for 6 months. The control subject group will also make visits to the endocrinologist every 3 months with laboratory test of A1c and serum creatinine measurements at 3-month intervals for 6 months.

The Intervention group will also receive standard care and will be asked to perform self-blood glucose monitoring 3 times daily for 6 months. However, the Intervention group will also be asked to report their blood glucose reading every 2 weeks through an Internet based glucose monitoring system. The Intervention group will also make visits to the endocrinologist every 3 months with A1c and serum creatinine measurements at 3-month intervals for 6 months. The laboratory measurements of both groups will be recorded and used for data analysis.

Statistical Analysis: The primary endpoint is the A1c level or the change in A1c level. The secondary endpoints include severe hypoglycemia defined as requiring external aid, hospital admissions for any CVD related intervention, and adverse events such as unplanned hospitalizations for any cause that last more than 24 hours. Patients who do not have the required number of SBGM tests performed or patients requiring new laser therapy will be asked to discontinue the study.

For each group, A1C levels before the start of study will be compared to A1C levels 3 and 6 months after the start of the study. Paired t-tests and random effects models (longitudinal analyses) will examine differences in A1C values before and after the study duration. Unpaired, independent t-tests will be done to examine the difference in A1C values between the two groups before and after the interventions. The planned sample size is 50.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients treated with insulin
* A1C 7-11%
* >25 years of age
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be randomized
* Trained in self blood glucose monitoring
* Internet Access

Exclusion Criteria:

* Patients who do not meet the inclusion criteria or are not willing to participate will not be included in the study.
* In addition patients with the potential to become pregnant or patients using medications known to influence control of diabetes (eg steroids systemic or inhaled) are excluded from the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the A1c level or the change in A1c level. | 6 months

SECONDARY OUTCOMES:
The secondary endpoints include severe hypoglycemia defined as requiring external aid, hospital admissions for any CVD related intervention, and adverse events such as unplanned hospitalizations for any cause that last more than 24 hours. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh D Tildesley, MD, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Karter AJ, Ackerson LM, Darbinian JA, D'Agostino RB Jr, Ferrara A, Liu J, Selby JV. Self-monitoring of blood glucose levels and glycemic control: the Northern California Kaiser Permanente Diabetes registry. Am J Med. 2001 Jul;111(1):1-9. doi: 10.1016/s0002-9343(01)00742-2. PMID 11448654
- [Derived] Tildesley HD, Mazanderani AB, Ross SA. Effect of Internet therapeutic intervention on A1C levels in patients with type 2 diabetes treated with insulin. Diabetes Care. 2010 Aug;33(8):1738-40. doi: 10.2337/dc09-2256. PMID 20668152